CLINICAL TRIAL: NCT05534334
Title: Corticosteroid Intralesional Injection as an Alternative Treatment in Oral Pyogenic Granuloma in the Esthetic Zone
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Eman Magdy Ahmed, Principal Investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17/4/21
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Oral Pyogenic Granuloma
MeSH Terms: interventions — hydrocortisone hemisuccinate; Hydrocortisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Active Comparator): Surgical excision of the gingival pyogenic granuloma
  Interventions: Drug: Solu-Cortef
- Intervention (Experimental): Intralesional injection with corticosteroids solution (1.8 mL of 100 mg hydrocortisone)
  Interventions: Drug: Solu-Cortef

INTERVENTIONS:
Drug: Solu-Cortef — A vial sol. used for intra-mascular injection
  Other Names: Hydrocortisone

SUMMARY:
Gingival Pyogenic granuloma in the esthetic zone represents an esthetic problem. While surgical treatment may not give the premium esthetic demands, corticosteroid may acheive this balance.

DETAILED DESCRIPTION:
In our practice, the investigators have found the use of topical steroids effectively induced regression of PGs. This protocol has been suggested by published case reports supported by the anti-inflammatory actions corticosteroid.

This is a particularly valuable approach for patients who have PG in the esthetic zone allowing the surgeon to keep maximum amount of periodontal tissues.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oral pyogenic granuloma at the esthetic zone

Exclusion Criteria:

* Patients who were not compliant to oral hygiene instructions and can not be motivated

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-29 (Estimated); Study Completion 2022-11-29 (Estimated)

PRIMARY OUTCOMES:
Remaining width of the attached gingiva | 6 month
  Remaining width of the attached gingival it is measured using graduated probe

SECONDARY OUTCOMES:
Recurrence of the lesion | 6 months
  Assessed as clinical reoccurrence of the lesion at the same site

CONTACTS AND LOCATIONS:
Overall Officials: Eman Magdy, PhD, Principal Investigator — Lecturer
Locations (2):
- Egypt (2):
  - Beni_Suef University, Banī Suwayf, Beni Suweif Governorate
  - Eman Ahmed, Banī Suwayf, Benisuef

IPD SHARING:
Plan to Share IPD: No